CLINICAL TRIAL: NCT04305899
Title: An Open-Label Cross-Over Study to Compare Bioavailability, Dose Proportionality, and Palatability of Single Doses of BMS-986165 Minitablet Pediatric Formulation in Fasted and Fed Conditions Relative to Single Doses of BMS-986165 Clinical Formulations In Healthy Adult Participants
Brief Title: A Study to Compare the Taste and Levels in Blood Plasma of BMS-986165 When Taken as Different Formulations by Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-113
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Treatment Group 1 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 2 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 3 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 4 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 5 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 6 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 7 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 8 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 9 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2
- Treatment Group 10 (Experimental)
  Interventions: Drug: BMS-986165 Tablet formulation 1; Drug: BMS-986165 Tablet formulation 2

INTERVENTIONS:
Drug: BMS-986165 Tablet formulation 1 — Specified dose on specified days
Drug: BMS-986165 Tablet formulation 2 — Specified dose on specified days

SUMMARY:
The purpose of this study is to compare the taste, and the levels in blood plasma of different tablet formulations of BMS-986165 when taken by healthy adults.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations in the opinion of the investigator
* Women and men must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of/or active liver disease
* Inability to tolerate oral medication
* History of allergy to BMS-986165 or related compounds

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) in plasma for BMS-986165 | Up to 26 days
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-T)) in plasma for BMS-986165 | Up to 26 days
Area under the plasma concentration-time curve extrapolated to infinity (AUC(INF)) in plasma for BMS-986165 | Up to 26 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 26 days
Incidence of Serious Adverse Events (SAEs) | Up to 98 days
Incidence of clinically significant changes in physical examination findings | Up to 68 days
Incidence of clinically significant changes in vital signs: Weight | Up to 68 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 68 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 68 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 68 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 68 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters | Up to 68 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 68 days
Incidence of clinically significant changes in clinical laboratory results: Clinical chemistry tests | Up to 68 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 68 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm